CLINICAL TRIAL: NCT00264264
Title: Arterial Closure vs Direct Compression for Hemostasis After Percutaneous Coronary Interventions
Brief Title: Arterial Closure vs Direct Compression for Hemostasis After PCI - The ACDC Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-101
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Angioplasty; Coronary Artery Disease
Keywords: Closure device; Stenting; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Vascular Closure Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Direct Compression (Active Comparator)
  Interventions: Procedure: Direct Compression
- Closure Device (Active Comparator)
  Interventions: Procedure: Closure Device

INTERVENTIONS:
Procedure: Closure Device
  Arms: Closure Device
Procedure: Direct Compression
  Arms: Direct Compression

SUMMARY:
Hemostasis at the arterial puncture site after percutaneous coronary interventions is achieved by either placement of a puncture closure device or by delaying sheath removal for hours to allow normalization of heparin induced anticoagulation. Both of these methods are far from ideal. Delayed sheath removal poses a risk of recurrent bleeding, hematoma formation and results in decreased patient mobility while the safety of closure devices has been called into question by several recent reports. Due to the lack of definitive data, the arterial access site management varies considerably between physicians and among institutions. The proposed study will evaluate the safety and efficacy of arterial closure devices to achieve hemostasis compared with immediate sheath removal after protamine administration followed by direct compression after percutaneous coronary intervention procedures.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the most common procedure performed for obstructive coronary artery disease with more than one million procedures performed annually in United States alone1. Despite major advances in technology and operative expertise, the optimum management of arterial access site after PCI procedures remains unclear.

The conventional practice of arterial access site management involves delaying of sheath removal for several hours to allow normalization of heparin induced anticoagulation. This delayed sheath removal poses a risk of recurrent bleeding and hematoma formation. Furthermore, delayed sheath removal results in decreased patient mobility, increased patient discomfort and requires frequent monitoring with an impact on nursing resources. The risks associated with delayed sheath removal may be further increased by concomitant administration of potent anti platelet therapy now routinely used in patients undergoing PCI2.

Arterial puncture closure devices (APCD) were developed to obtain immediate arterial access site hemostasis after closed vascular procedures with an aim towards early patient mobilization. Although the efficacy of APCD have been documented in several small studies but limited information is available regarding their safety in diverse patient populations. A recent meta analysis has shown increased vascular complication rate associated with the use of these devices bringing the safety of their routine use into question3.

Due to lack of definitive data, the arterial access site management varies considerably between physicians and among institutions. APCD are routinely used by some centers4 while others continue to delay arterial sheath removal for several hours after the procedure5.

Immediate sheath removal followed by direct compression though routinely practiced after coronary angiographic procedures is not used after PCI procedures due to the intra procedural administration of heparin resulting in prolonged anticoagulation. Reversal of heparin with protamine may allow immediate sheath removal resulting in early patient ambulation and decreased access site vascular complications. The safety and efficacy of intravenous protamine administration for reversal of heparin is well established by its routine use in cardiovascular surgery for several decades6 and recent reports showing safety and efficacy of this method for early sheath removal after PCI procedures7-9.

The proposed study is designed to evaluate the safety and efficacy of immediate sheath removal followed by direct compression as compared to the use of APCD to achieve hemostasis after PCI.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective PCI procedures. Femoral artery anatomy favorable for the placement of a closure device Planned use of clopidogrel and platelet glycoprotein IIb/IIIa antagonist

Exclusion Criteria:

Emergency PCI End stage renal disease Hemoglobin level < 100g/l Fish Allergy. Known allergy to Protamine. Use of low molecular weight heparin within last 12 hours. Prior closure device use within 90 days. Symptomatic peripheral vascular disease. Femoral artery calcification on fluoroscopy. Arterial puncture of the superficial femoral artery. Double wall puncture (puncture of anterior & posterior wall of femoral artery). Placement of intra aortic balloon pump. Placement of a femoral venous sheath. Coronary dissection, thrombus or perforation not resolved by the end of case

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2006-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
A composite of major vascular complications (device failure, bleeding, hematoma, infection, pseudoaneurysm, AV fistula and vascular repair)

SECONDARY OUTCOMES:
Time to hemostasis
Ambulation time
Quality of life
Composite of minor vascular complication (bleeding, repeat compression, failure to ambulate per protocol),
Post procedural infarction
30 day MACE (death, MI, TVR)

CONTACTS AND LOCATIONS:
Overall Officials: Asim Cheema, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada